CLINICAL TRIAL: NCT01378663
Title: Review of Pain Management After Congenital Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Aymen N Naguib, Director of Pediatric Cardiothoracic Anesthesia, Nationwide Children's Hospital
Other Study IDs: IRB10-00058
Record Dates: First submitted 2011-06-21; First posted 2011-06-22 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Postoperative Pain Management
Keywords: Congenital cardiac surgery; Postoperative pain management

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Post congenital cardiac surgery pain management: All patients that underwent congenital cardiac surgery from 2004 till 2010 and required PCA or NCA.

SUMMARY:
One of the main problems that faces children undergoing congenital cardiac surgery is posoperative pain management. PCAs (Patient Controlled Analgesia) and NCAs (Nurse Controlled Analgesia) are the main means of pain management here at NCH. In this study, the investigators will review the difference between different PCA and NCA modalities. Also, the investigators aim to find out if there are differences between age groups in terms of type of drug used, total drug used, side effects and length of use of the PCA or NCA.

DETAILED DESCRIPTION:
All patients that underwent congenital cardiac surgery from 2004 till 2010 and required PCA or NCA will be included. Data will be collected from the pain team database and charts review. Data will include; patient's age, weight, sex, procedure, pain scores and sedation score during the times of PCA and NCA use, side effects (respiratory depression, nausea, vomitting, pruritus, itching and other).In addition we will record the total days of PCA and NCA use. We will also look at the incidence of changes done in the PCA/NCA and drug itself.

Identifying the ideal drug and dose based on the patient's age and procedure will allow us to take better care of our patients. Our patient population is peculiar in the fact that a big percentage of our patients are extubated in the Operating Room. For this reason, sedation and analgesia play an important role for our continued success in taking care of them.

ELIGIBILITY:
Inclusion Criteria:

* All patients that underwent congenital cardiac surgery from 2004 till 2010 and required PCA or NCA.

Exclusion Criteria:

* All patients that underwent congenital cardiac surgery from 2004 till 2010 and did not receive PCA or NCA for postoperative pain management.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients that underwent congenital cardiac surgery from 2004 till 2010 and required PCA or NCA.
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aymen N Naguib, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Howard RF, Lloyd-Thomas A, Thomas M, Williams DG, Saul R, Bruce E, Peters J. Nurse-controlled analgesia (NCA) following major surgery in 10,000 patients in a children's hospital. Paediatr Anaesth. 2010 Feb;20(2):126-34. doi: 10.1111/j.1460-9592.2009.03242.x. PMID 20078810